CLINICAL TRIAL: NCT03857789
Title: Supporting Health Care Professionals With a Social Robot in an Integrated Care Pathway: A Randomized Controlled Trial
Brief Title: Social Robot Support for Healthcare Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Delft University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2018-5019
Record Dates: First submitted 2019-02-15; First posted 2019-02-28 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2019-02

CONDITIONS: Frailty at Older Adults
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular care (Other): Participant will be received by Healthcare professional (HCP). The HCP will administer a questionnaire. The HCP will discuss the results.
  Interventions: Other: Questionnaire
- New care (Experimental): Participant will be received by Healthcare professional (HCP). The social robot will administer a questionnaire. The HCP will discuss the results.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A 40 question frailty questionnaire.

SUMMARY:
This study evaluates the effectiveness of integrated care pathway steps supported by social robots. Half of the participants will receive regular care, while for the other half a social robot dialogue will be included as part of the pathway step.

DETAILED DESCRIPTION:
There is a worldwide increasing shortage of adequately trained healthcare personnel, leading to the challenge for society to prevent a future "lack of care". At the same time the number of people requiring healthcare is expanding rapidly, amongst others due to the growing percentage of older adults in the population. New means of supporting the available healthcare professionals are therefore urgently required.

Modern healthcare is often implemented through "integrated care pathways". Certain steps in these pathways involve dialogues with patients. Speaking social robots are increasingly being advertised as supportive for healthcare professionals and may handle certain structured dialogue types, such as questionnaires. Based on previous positive preclinical experiences with social robots interviewing community-dwelling older subjects, the researchers want to investigate the implementation of a social robot in an integrated care pathway in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of need for quality of life support

Exclusion Criteria:

* Psychiatric Disorders

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Consumer Quality index (CQ-index) | 4 Months
  The CQ-index records the quality of care from a patient perspective using answers to questions like "Would you recommend this outpatient clinic to your family?", "How did you experience the communication with your caregiver?" and "Were you adequately informed?".

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boumans R, van Meulen F, van Aalst W, Albers J, Janssen M, Peters-Kop M, Huisman-de Waal G, van de Poll A, Hindriks K, Neerincx M, Olde Rikkert M. Quality of Care Perceived by Older Patients and Caregivers in Integrated Care Pathways With Interviewing Assistance From a Social Robot: Noninferiority Randomized Controlled Trial. J Med Internet Res. 2020 Sep 9;22(9):e18787. doi: 10.2196/18787. PMID 32902387